CLINICAL TRIAL: NCT05385523
Title: Comparison Between Analgesic Effect of Adding Dexamedatomidine or Dexamethasone to Bupvicaine in Rhomboidal Intercostal Plain Block and Subserratus Block in Breast Surgery
Brief Title: Dexamedatomidine vs. Dexamethasone in Rhomboidal Intercostal Plain Block and Subserratus Block in Breast Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Armed Forces College of Medicine, Cairo, Egypt (Other)
Responsible Party: Principal Investigator, bassant mohamed, Professor, Armed Forces College of Medicine, Cairo, Egypt
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 97
Record Dates: First submitted 2022-05-18; First posted 2022-05-23 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2022-05

CONDITIONS: Postoperative Pain, Acute
MeSH Terms: conditions — Pain, Postoperative | interventions — Anesthesia, General; Dexamethasone; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- dexamedatomidine (Experimental): Patients will receive general anaesthesia and RISS block with 20 ml of 0.25% bupivacaine + 1 Mcg/kg dexamedatomidine in 2 mL.
  Interventions: Procedure: Rhomboid Intercostal and Sub-Serratus block technique (RISS); Procedure: General Anaesthesia; Drug: dexamedatomidine
- dexamethasone (Experimental): Patients will receive general anaesthesia and RISS block with 20 ml of 0.25% bupivacaine + 8mg dexamethasone in 2 mL.
  Interventions: Procedure: Rhomboid Intercostal and Sub-Serratus block technique (RISS); Procedure: General Anaesthesia; Drug: dexamethasone
- saline (Experimental): Patients will receive general anaesthesia and RISS block with 20 ml of 0.25% bupivacaine+ 2 mL normal saline.
  Interventions: Procedure: Rhomboid Intercostal and Sub-Serratus block technique (RISS); Procedure: General Anaesthesia; Drug: saline

INTERVENTIONS:
Procedure: Rhomboid Intercostal and Sub-Serratus block technique (RISS) — The patient will be placed in lateral position. A linear ultrasound transducer of frequency 6-12 MHz will be placed medial to the lower border of the scapula in a sagittal plane. A 38-mm 22-gauge will be inserted under real-time in-plane from craniocaudal between the rhomboid major and intercostal muscles. After negative aspiration, single injection of 10 ml of the local anesthetic mixture will be administered at the T6 7 level. The spread of local anesthetic solution under the rhomboid muscle will be visualized by ultrasonography. Then the ultrasound probe will be moved caudally and laterally to identify the tissue plane between the serratus anterior and external intercostal muscle for the sub-serratus block at T 8-9 level. The needle will be advanced from its previous position and a further of 10 ml of the local anesthetic mixture will be injected.
Procedure: General Anaesthesia — Fentanyl (1 μg/kg), propofol (2-3mg/kg) and atracurium (0.3-0.5 mg/kg) will be injected intravenously 3-5 minutes after oxygenation. A single-lumen endotracheal tube will be used to complete ventilation. The ventilator ventilation mode is volume control mode, and the patient's end-expiratory carbon dioxide level is maintained at 35-40 mmHg throughout the anesthesia process. During the anesthesia maintenance phase, 2% sevoflurane mixed with 60% oxygen.
  After general anaesthesia induction, all patients will receive RISS block with different local anesthetic drug mixture according to randomization.
Drug: dexamedatomidine — Patients will receive general anaesthesia and RISS block with 20 ml of 0.25% bupivacaine + 1 Mcg/kg dexamedatomidine in 2 mL.
  Arms: dexamedatomidine
Drug: dexamethasone — Patients will receive general anaesthesia and RISS block with 20 ml of 0.25% bupivacaine + 8mg dexamethasone in 2 mL.
  Arms: dexamethasone
Drug: saline — Patients will receive general anaesthesia and RISS block with 20 ml of 0.25% bupivacaine+ 2 mL normal saline.
  Arms: saline

SUMMARY:
The aim of this study is to evaluate the analgesic efficacy and safety of adding dexmedetomidine and dexamethasone to bupivacaine in rhomboidal intercostal and subserratus (RISS) block for patients undergoing modified radical mastectomy compared to bupivacaine only.

DETAILED DESCRIPTION:
Rhomboid intercostal block (RIB); a new interfascial plane block involves the triangle of auscultation that's bounded medially by inferior a part of the trapezius, inferiorly by the superior border of latissimus dorsi, and laterally by the medial border of the scapula. The local anaesthetic spreads between the rhomboid major and therefore the intercostal fascia at the extent of T6-T7 and provides analgesia of T3-T8 dermatomes.

Aiming to expand dermatomal coverage, a new modification of Rhomboid Intercostal and Sub-Serratus block (RISS) is performed by advancing the ultrasound probe caudally and laterally distal to the inferior angle of the scapula, the second injection apply between the serratus and intercostal muscle fascia. The RISS block is a novel ultrasound-guided block that has been shown to provide analgesia from T2-T11 dermatomes.

Dexmedetomidine is a potent selective α 2 adrenoceptor agonist that was reported in many previous studies as an adjunct to regional and general anesthesia, with significant prolongation of the duration of sensory block, motor block and analgesia, and accelerate the time to onset of sensory and motor block when added to a local anesthetic.

Dexamethasone is a potent long-acting steroid that has shown efficacy as an adjuvant to local anesthetics in various studies. It enhances peripheral nerve blocks when added to local anesthetics, providing better quality of anesthesia as well as postoperative analgesia. The mechanism by which dexamethasone prolong the duration of local anesthetics are not completely understood; however, some studies demonstrated that dexamethasone exerts its action through reducing the release of inflammatory mediators and by inhibiting discharge of C-fibers.

ELIGIBILITY:
Inclusion Criteria:

* Adult female patient
* Type of surgery; Modified Radical Mastectomy (MRM).
* Physical status ASA II, III.
* Age ≥ 21 and ≤ 65 Years.
* Body mass index (BMI): > 20 kg/m2 and < 35 kg/m2.

Exclusion Criteria:

* Patient refusal.
* Patients suffering from coagulation disorders.
* Patients with histories of allergic reactions to local anesthetics or dexmedetomidine.
* Patients suffering from neuropsychiatric disorders.
* Pregnancy.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-07-20 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Time of first request of analgesia. | 24 hours
  calculated from the time of complete injection of local anesthetics till the numerical rating scale (is more than or equals 3

SECONDARY OUTCOMES:
Total amount of morphine consumption | 24 hours
mean arterial blood pressure | 24 hours
heart rate | 24 hours
Numerical rating scale | 24 hours
  The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").

CONTACTS AND LOCATIONS:
Overall Officials: Bassant Abdelhamid, MD, Principal Investigator — AFCM Egypt
Locations (1):
- AFCM Egypt, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Elsharkawy H, Ince I, Pawa A. Rhomboid intercostal and sub-serratus (RISS) plane block for analgesia after lung transplant. J Clin Anesth. 2019 Sep;56:85-87. doi: 10.1016/j.jclinane.2019.01.042. Epub 2019 Jan 28. No abstract available. PMID 30703673
- [Background] Kaur H, Singh G, Rani S, Gupta KK, Kumar M, Rajpal AS, Aggarwal S. Effect of dexmedetomidine as an adjuvant to levobupivacaine in supraclavicular brachial plexus block: A randomized double-blind prospective study. J Anaesthesiol Clin Pharmacol. 2015 Jul-Sep;31(3):333-8. doi: 10.4103/0970-9185.161668. PMID 26330711
- [Background] Bjorn S, Linde F, Nielsen KK, Borglum J, Hauritz RW, Bendtsen TF. Effect of Perineural Dexamethasone on the Duration of Single Injection Saphenous Nerve Block for Analgesia After Major Ankle Surgery: A Randomized, Controlled Study. Reg Anesth Pain Med. 2017 Mar/Apr;42(2):210-216. doi: 10.1097/AAP.0000000000000538. PMID 28033159